CLINICAL TRIAL: NCT01108770
Title: Evaluation of Phenotypic and Genetic Properties in Male Subjects With Hypohidrotic Ectodermal Dysplasia and Their Family Members
Brief Title: Evaluation of Phenotypic and Genetic Properties in Male Subjects Affected By Hypohidrotic Ectodermal Dysplasia
Status: Completed | Type: Observational
Sponsor: Edimer Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: ECP-001
Record Dates: First submitted 2010-04-21; First posted 2010-04-22 (Estimated); Last update posted 2012-08-21 (Estimated); Status verified 2012-08

CONDITIONS: Ectodermal Dysplasia
Keywords: HED; XLHED; Hypohidrotic Ectodermal Dysplasia
MeSH Terms: conditions — Ectodermal Dysplasia; Ectodermal Dysplasia 1, Anhidrotic

STUDY DESIGN:
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HED affected males
- Unaffected male controls

SUMMARY:
To characterize skin properties in male subjects with HED

DETAILED DESCRIPTION:
This study is designed to obtain information from male subjects with HED and unaffected male control subjects. The study will consist of the standardized collection of data from HED medical history questionnaires and non-invasive tests. A subset of subjects will undergo genetic testing. All data will be collected from families attending the 2010 NFED Family Conference, July 22-24, 2010, in Colorado Springs, CO.

Since HED is a rare disease, it is difficult to obtain reliable data on a sufficient number of subjects in any one region. The NFED Family Conference is a location where families affected with HED come together, and therefore, presents an ideal location to obtain data needed to design future studies. As the procedures are non-invasive and are designed to take a relatively short period of time, subjects can participate in this study while attending the NFED Family Conference.

ELIGIBILITY:
Inclusion Criteria:

1. Registered and attending the 2010 NFED Family Conference;
2. One year of age or greater;
3. Conform to one of the following requirements for providing informed consent:

   * if more than 18 years of age, subjects must provide signed informed consent;
   * if less than 18 years of age and it is determined that the subject is capable of providing assent, both the assent of the subject and consent of the parent(s) or guardian of that subject must be granted. Under this condition, both parents of the subject should give their permission, unless 1 parent is deceased, unknown, incompetent, or not available;
   * if the subject is incapable of providing assent, the consent of the parent(s) or guardian of the subject must be granted. Under this condition, both parents should give their consent, unless 1 parent is deceased, unknown, incompetent, or not available.
4. Subjects must meet one of the following criteria:

   * Male subjects of original gender with the clinical characteristics of HED, including at least a history of decreased sweating and either abnormal teeth (fewer permanent teeth, teeth are smaller than average and often have conical crowns), and/or sparseness of scalp and body hair;
   * Healthy male controls, i.e. either unaffected male family members or unaffected male volunteers.

Exclusion Criteria:

1. Known hypersensitivity to pilocarpine or pilocarpine-like muscarinic agonists.
2. Presence of pacemakers.
3. Subjects who are not able or are not willing to comply with the procedures of this protocol.
4. Subjects with any major medical problem that will prevent them from participating in this study.

Min Age: 1 Year | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Male subjects with HED or unaffected controls
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2010-07; Primary Completion 2010-07 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Characterization of skin properties in HED affected male subjects compared with healthy controls | Two assessments conducted once during study day.
  The primary objective of this descriptive study is to use skin assessment techniques to characterize skin properties in male subjects affected by HED compared with healthy controls including determination of the number of sweat glands and the rate of sweating.

SECONDARY OUTCOMES:
Collecting demographic information and clinical status in male subjects affected by HED using a medical questionnaire. | Collected once during study day.
Testing for the presence of ectodysplasin A (EDA) gene mutations in a subset of subjects enrolled in this study. | Collected once during study day.

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy K Grange, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Cheyenne Mountain Resort, Colorado Springs, Colorado, United States